CLINICAL TRIAL: NCT02692391
Title: A Randomized Controlled Pilot Trial of Indomethacin in Acute Pancreatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, David Whitcomb, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY19050212
Record Dates: First submitted 2016-02-15; First posted 2016-02-26 (Estimated); Results first posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-03

CONDITIONS: Acute Pancreatitis
Keywords: Acute pancreatitis; Indomethacin; Organ failure; Prevention
MeSH Terms: conditions — Pancreatitis | interventions — Indomethacin; Glycerol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): 6 doses, Q8hrs for a total period of 48 hours
  Interventions: Drug: Placebo
- Indomethacin suppository (Active Comparator): Loading dose :100mg Maintenance dose: 50 mg, Q8hrs for a total period of 48 hours (5 doses)
  Interventions: Drug: Indomethacin

INTERVENTIONS:
Drug: Indomethacin — Rectal indomethacin will be administered as 100 mg loading doses following by 5 maintenance doses of 50 mg at internals of 8 hours for total of 48 hours.
  Other Names: Indocin
  Arms: Indomethacin suppository
Drug: Placebo — Glycerin placebo suppositories which are identical in shape, size, color, and packaging to rectal indomethacin
  Other Names: Glycerin
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled pilot trial seeking to evaluate the efficacy of rectal indomethacin in abrogating systemic inflammation and subsequently organ failure and mortality in patients with AP and positive SIRS score.

DETAILED DESCRIPTION:
Background:

AP is an inflammatory disease with a highly variable clinical course that is potentially lethal. This disease is currently the leading cause of gastrointestinal-related hospital admissions in the United States and continues to rise in incidence. The inciting event leading to the development of AP is the premature activation of the digestive pro-enzyme trypsinogen to trypsin within pancreatic acinar cells, resulting in pancreatic auto-digestion and inflammation. Inflammation localized to the gland can subsequently progress to a systemic inflammatory response affecting distant organs.

Studies have revealed a key role for phospholipase A2 in propagating this inflammatory response by inducing the production of inflammatory mediators, including arachidonic acid metabolites. Elevated levels of phospholipase A2 have been found in the serum of patients with AP who develop severe complications, including pancreatic necrosis, shock, and OF. The in vitro inhibition of phospholipase A2 using NSAIDs has been evaluated as a potential treatment strategy for AP, with indomethacin shown to be the most potent inhibitor among 17 tested agents. NSAIDs also inhibit the interaction of neutrophils with endothelial cells, thus preventing the accumulation of neutrophils at the site of injury.

In animal models of AP, NSAIDs have been shown to attenuate AP severity and improve survival. Most human studies, however, have primarily assessed the role of NSAIDs in PEP prophylaxis. A meta-analysis of 4 randomized, controlled studies evaluating this effect revealed a protective role for these medications, and a recent multicenter, randomized controlled trial found that administrating rectal indomethacin to patients at increased risk for PEP significantly reduced the incidence and severity of pancreatitis. In 1985, a small randomized controlled trial (n=30) of rectal indomethacin in patients with AP reported a significant decrease in the duration of pain. This is the only study to date evaluating NSAIDs following the onset of AP and did not evaluate systemic inflammation. The effect of rectal indomethacin in mitigating disease progression in patients at risk for developing severe disease thus remains to be evaluated.

SIRS is a simple clinical score, ranging from 0-4, that utilizes objective, routine clinical parameters (body temperature, heart rate, respiratory rate or arterial carbon dioxide tension and white blood count) that directly reflect the underlying inflammatory response. The persistence of SIRS, defined by the presence of a SIRS score ≥2 at 48 hrs following presentation, has been shown to be significantly associated with the development of OF, pancreatic necrosis and death in patients with AP. Additionally, serum levels of CRP at 48 hours following admission have also been closely correlated with the development of OF.

Objective:

Our proposed randomized, double-blind, placebo-controlled pilot trial seeks to evaluate the efficacy of rectal indomethacin in abrogating systemic inflammation in patients with acute pancreatitis (AP) and systemic inflammatory response syndrome (SIRS).

Specific Aims:

Our long-term goal is to alter the clinical course of AP in patients who are at high risk for the development of organ failure (OF) and death. The objective of this randomized, double-blind, placebo-controlled pilot trial is to evaluate the efficacy of rectal indomethacin on attenuating systemic inflammation in patients with AP who also have SIRS. The investigators hypothesize that the treatment of patients with AP and SIRS with therapeutic doses of rectal indomethacin will mitigate the inflammatory response through the inhibition of inflammatory mediators. The investigators will also test the hypothesis by enrolling 42 patients randomized to receive either rectal indomethacin or placebo for 48 hours and pursuing the following specific aims:

Aim 1. Evaluate the effect of rectal indomethacin on systemic inflammation as measured by the change in mean SIRS score and serum CRP levels following 48hrs of treatment in patients with AP and SIRS; and

Aim 2. Evaluate the impact of rectal indomethacin on the development of OF and mortality.

Significance:

The proposed study will thus be the first attempt at evaluating the therapeutic role of NSAIDs in patients with AP and SIRS who are at high risk for the development of OF and for whom no effective pharmacological therapy is currently available. Pilot data generated will serve as a platform for a larger scale study that will validate the efficacy of indomethacin in the treatment of AP.

ELIGIBILITY:
Inclusion Criteria:

* All patients ages 18 or above admitted to UPMC with a diagnosis of AP based on at least 2 of the following criteria:

  (i) abdominal pain characteristic of AP (ii) serum amylase and/or lipase ≥ 3 times the upper limit of normal (iii) characteristic findings of AP on abdominal CT scan will be screened for study enrollment.
* Patients with SIRS (≥ 2 of the following criteria: temperature <36°C or >38°C, heart rate >90/min, respiratory rate >20/min OR PaCO2<32 mmHg, WBC <4,000/mm3, >12,000/mm3 or >10% bands) upon hospital admission or who develop SIRS during their first week of hospitalization

Exclusion Criteria:

* Presence of OF (shock defined by SBP<90mmHg, PO2<60mmHg on room air or need for mechanical ventilation, Cr≥2mg/dL)
* Presence of renal dysfunction (Cr>1.5mg/dL)
* Active peptic ulcer disease
* Pregnancy
* Use of daily NSAIDs within 1 week of presentation
* Allergy to NSAIDs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georgios I Papachristou, MD PhD, Study Chair — Ohio State University
Locations (1):
- Univeristy of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sotoudehmanesh R, Eloubeidi MA, Asgari AA, Farsinejad M, Khatibian M. A randomized trial of rectal indomethacin and sublingual nitrates to prevent post-ERCP pancreatitis. Am J Gastroenterol. 2014 Jun;109(6):903-9. doi: 10.1038/ajg.2014.9. Epub 2014 Feb 11. PMID 24513806
- [Result] Freeman ML, Guda NM. Prevention of post-ERCP pancreatitis: a comprehensive review. Gastrointest Endosc. 2004 Jun;59(7):845-64. doi: 10.1016/s0016-5107(04)00353-0. No abstract available. PMID 15173799
- [Derived] Machicado JD, Mounzer R, Paragomi P, Pothoulakis I, Hart PA, Conwell DL, de-Madaria E, Greer P, Yadav D, Whitcomb DC, Lee PJ, Hinton A, Papachristou GI. Rectal Indomethacin Does Not Mitigate the Systemic Inflammatory Response Syndrome in Acute Pancreatitis: A Randomized Trial. Clin Transl Gastroenterol. 2021 Oct 27;12(11):e00415. doi: 10.14309/ctg.0000000000000415. PMID 34704970

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Indomethacin Suppository
Started | 24 | 18
Completed | 24 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Indomethacin Suppository | Total
Number analyzed (Participants) | 24 | 18 | 42
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47.5 [35.6 to 63.1] | 50.8 [42.2 to 61.1] | 50.8 [37.2 to 62.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 16 | 7 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 18 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 20 | 15 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 18 | 42
BMI, continuous [Median (Inter-Quartile Range); unit: kg/m^2] | 31.7 [26.9 to 37.4] | 27.8 [23.1 to 35.2] | 30 [24.3 to 36.4]

OUTCOME MEASURES:

1. Primary Outcome: Systemic Inflammatory Response Syndrome (SIRS) Score
Description: SIRS is a simple clinical score, ranging from 0-4, that utilizes objective, routine clinical parameters (body temperature, heart rate, respiratory rate or arterial carbon dioxide tension and white blood count) that directly reflect the underlying inflammatory response. A lower change in SIRS score (negative number) indicates a better outcome (less inflammation).
Time Frame: The change in the SIRS score (48 hours - baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Indomethacin Suppository
Number analyzed (Participants) | 24 | 18
score on a scale | -0.96 (0.81) | -1 (1.24)
Statistical Analysis 1: Comparison: Placebo vs Indomethacin Suppository; Test type: Superiority; p = 0.87, Wilcoxon (Mann-Whitney)

2. Primary Outcome: C-Reactive Protein (CRP) Levels.
Description: CRP levels at 48 hours after enrollment minus CRP levels at enrollment (baseline). A negative number indicates a better outcome (less inflammation).
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Indomethacin Suppository
Number analyzed (Participants) | 24 | 18
mg/dL | -1.43 (8.73) | -2.08 (12.55)
Statistical Analysis 1: Comparison: Placebo vs Indomethacin Suppository; Test type: Superiority; p = 0.48, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Number of Participants Who Development of Organ Failure
Description: Including respiratory, renal and cardiovascular failures defined as modified Marshal score of equal and greater than 2. The minimum and maximum values in the modified Marshal score for each organ failure range from 0 to 4 with a higher value representing worse outcomes.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Indomethacin Suppository
Number analyzed (Participants) | 24 | 18
Participants | 6 | 3
Statistical Analysis 1: Comparison: Placebo vs Indomethacin Suppository; Test type: Superiority; p = 0.71, Fisher Exact

4. Secondary Outcome: Mortality
Description: Enrolled subjects that died. A death indicates a worse outcome.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Indomethacin Suppository
Number analyzed (Participants) | 24 | 18
Participants | 1 | 0
Statistical Analysis 1: Comparison: Placebo vs Indomethacin Suppository; Test type: Superiority; p = 1.00, Fisher Exact

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Placebo | Indomethacin Suppository
All-Cause Mortality (participants affected / at risk) | 1/24 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/18
Other Adverse Events (participants affected / at risk) | 2/24 | 0/18
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | Indomethacin Suppository (N=18)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
GI Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2013-06-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT02692391/Prot_000.pdf
  • Statistical Analysis Plan (2013-06-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT02692391/SAP_001.pdf